CLINICAL TRIAL: NCT06684600
Title: A Single-arm, Phase II Clinical Trial of Dalpiciclib Combined with Pyrotinib As Second-line Treatment of Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Study of Dalpiciclib Isethionate Plus Pyrotinib Maleate in the Treatment of Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024YJZ118
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — dalpiciclib; pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dalpiciclib + Pyrotinib (Experimental)
  Interventions: Drug: Dalpiciclib + Pyrotinib

INTERVENTIONS:
Drug: Dalpiciclib + Pyrotinib — Dalpiciclib Isethionate tablets, 125mg, oral administration on days 1 to 21, followed by a 7-day drug holiday, every 4 weeks; Pyrotinib Maleate tablets, 320mg, oral administration once daily on days 1 to 28, every 4 weeks; Treatment will continue until disease progression, intolerable toxicity, initiation of new antitumor therapy, withdrawal of informed consent, or the investigator determines that the subject should discontinue study treatment.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of dalpiciclib combined with pyrotinib as second-line therapy in patients with advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The incidence of esophageal cancer is ranked seventh in the world, and the mortality rate ranks sixth in the world. At present, the first-line treatment of advanced esophageal cancer is mainly based on the combination of paclitaxel, cisplatin and fluorouracil. After the failure of first-line treatment, there is no standard second-line treatment. The investigators designed a single-arm, phase II clinical trial of dalpiciclib combined with pyrotinib as second-line therapy in patients with advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18~75 years, both men and women.；
2. Pathologically (histologically or cytologically) confirmed diagnosis of esophageal squamous cell carcinoma (ESCC), and local recurrence or distant metastasis；
3. Patients undergoing first-line systemic chemotherapy progression or intolerance (progress in maintenance therapy after first-line chemotherapy can also be included). Synchronous chemoradiotherapy for postoperative recurrence or metastasis is considered as first-line treatment; For radical concurrent chemoradiotherapy, neoadjuvant/adjuvant therapy (chemotherapy or chemoradiotherapy), if disease progression occurs during treatment or within 6 months after stopping treatment, Count it as a first-line treatment failure.
4. At least one measurable/evaluable lesion by RECIST v1.1. And the measurable lesions should not have received local treatment such as radiotherapy (The lesion located in the previous radiotherapy area, if confirmed to progress, and meets the RECIST 1.1 standard, can also be used as a target lesion).
5. Tissue samples shall be provided for biomarker analysis, preferably newly acquired tissues, and patients who are unable to provide newly acquired tissues may provide 5-8 pieces of 5um thick paraffin sections that are archived and preserved.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Capable of swallowing tablets normally.
8. Life expectancy of ≥ 12 weeks.
9. The main organs function normally, that is, the following criteria are met:

   1. ANC≥1.5×109/L
   2. PLT≥90×109/L；
   3. HB≥90g/L；
   4. ALB≥28g/L；
   5. TBIL≤1.5 × ULN，ALT and AST ≤ 2.5ULN; if there is liver metastasis, ALT and AST ≤ 5ULN
   6. plasma Cr ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min.
   7. APTT and INR ≤1.5 × ULN
10. Female subjects of childbearing potential must undergo a blood pregnancy test within 72 hours prior to the first administration of the drug and the result must be negative. They must not be breastfeeding and must agree to use effective contraception during the trial period and for at least 7 months after the last use of Dalpiciclib or at least 8 weeks after the last use of Pyrotinib, whichever is longer. Male subjects with partners of childbearing potential must be surgically sterilized or agree to use effective contraception during the trial period and for at least 7 months after the last use of Dalpiciclib or at least 8 weeks after the last use of Pyrotinib, whichever is longer. Sperm donation is not allowed during the study period.
11. Subjects voluntarily joined the study, signed informed consent, and were well-adhered to follow-u.

Exclusion Criteria:

1. Presence of clinically significant symptoms and uncontrollable third-space fluid accumulations, such as large pleural effusions or ascites, that cannot be managed through drainage or other methods.
2. Chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis) and intestinal obstruction, among other factors that may affect medication intake and absorption.
3. Prolonged corticosteroid therapy exceeding 30 days or requiring long-term corticosteroid use.
4. Prior radiotherapy, chemotherapy, hormonal therapy, surgery, or molecular-targeted therapy within 4 weeks of enrollment (eligible for enrollment if the last dose of anti-neoplastic medication was discontinued for ≥5 half-lives before the initial treatment); prior chemotherapy with nitrosoureas or mitomycin within 6 weeks of enrollment.
5. Unresolved adverse events related to prior treatments to less than grade 2 (excluding alopecia, asthenia, and adverse events deemed by the investigator not to affect eligibility).
6. Participation in another clinical trial of a new drug within 4 weeks, unless the trial is observational (non-interventional) or in a follow-up phase.
7. Persistent uncorrectable hypokalemia and hypomagnesemia at the time of enrollment.
8. Symptomatic or untreated brain metastases.
9. History of other malignancies within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
10. Concurrent administration of other anti-neoplastic treatments.
11. Individuals with an allergic constitution or known hypersensitivity to any component of the study medication.
12. Patients with a propensity for gastrointestinal bleeding, including but not limited to:

1) Active ulcers with fecal occult blood (++); 2) History of melena or hematemesis within the past 2 months; 3) For fecal occult blood (+) and the primary tumor site not surgically removed, a gastroscopy is required, and patients with visible active bleeding are ineligible.

13. Active infections, including but not limited to tuberculosis. 14. History of immunodeficiency, including positive HIV testing, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.

15. Severe cardiac conditions within the past 6 months, including but not limited to:

1. Acute coronary syndrome;
2. Clinically significant arrhythmias requiring medication or unable to discontinue medications that may prolong the QT interval during the study;
3. Acute myocardial infarction;
4. Heart failure;
5. Any other cardiac condition deemed unsuitable for trial participation by the investigator.

16. Pregnant or lactating women, or women of childbearing potential with a positive baseline pregnancy test.

17. Serious comorbidities judged by the investigator to endanger patient safety or impede study completion, such as hypertension, severe diabetes, thyroid disorders, etc.

18. Habitual alcohol consumption, smoking (≥5 cigarettes daily), and other detrimental lifestyle habits; heavy episodic drinking is defined as consuming approximately four or more drinks within 2 hours, where one drink is equivalent to 150 mL of wine, 350 mL of beer, or 50 mL of 80-proof spirits.

19. History of definite neurological or psychiatric disorders, including epilepsy or dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | an expected average of 24 months
  Proportion of subjects in the analysis population who achieved complete response (CR) or partial response (PR) based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival（OS） | an expected average of 24 months
  Time from initial treatment to the subject's death. At the end of the study, if the subject is still alive, the last known date of survival of the subject will be the date of deletion.
Progression-free Survival (PFS) | an expected average of 24 months
  Time from initial treatment to first radiographic disease progression (RECIST 1.1 criteria) or death, whichever occurs first.
Disease Control Rate (DCR) | an expected average of 24 months
  Proportion of subjects in the analysis population who achieved complete response (CR) , partial response (PR) or stable disease(SD) based on RECIST 1.1 criteria.
Adverse events | an expected average of 24 months
  The incidence and severity of adverse events (AE) and serious adverse events (SAE) were determined according to NCI-CTCAE v5.0 criteria.

OTHER OUTCOMES:
Correlations between biomarkers and clinical activity | an expected average of 24 months
  tumor biopsies are collected before start of treatment, for assessing the relationship between different biomarkers with Dalpiciclib and Pyrotinib regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihao Lu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Department of GI Oncology, Peking University Cancer Hospital,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No